CLINICAL TRIAL: NCT04050020
Title: The Effect of Platelet-rich Plasma(PRP) Injection Treatment on Erectile Function: a Double-blind, Placebo Controlled Randomized Clinical Trial
Brief Title: Platelet-rich Plasma (PRP) Injection for Treatment of Erectile Function
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Institute for the Study of Urological Diseases, Greece (Other)
Collaborators: European Society for Sexual Medicine (Unknown)
Responsible Party: Principal Investigator, Dimitrios Hatzichristou, Professor, Institute for the Study of Urological Diseases, Greece
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 65-08/10/18
Record Dates: First submitted 2019-08-06; First posted 2019-08-08 (Actual); Last update posted 2020-10-20 (Actual); Status verified 2020-10

CONDITIONS: Erectile Dysfunction Due to Arterial Insufficiency
Keywords: PRP; Platelet-Rich Plasma
MeSH Terms: interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator)
  Interventions: Biological: Platelet-Rich Plasma (PRP)
- Group B (Placebo Comparator)
  Interventions: Biological: Normal saline injection

INTERVENTIONS:
Biological: Platelet-Rich Plasma (PRP) — All subjects of this group will receive 2 sessions of PRP penile injection with 30 +/- 3 day treatment interval, 10 ml of PRP will be injected at each session.
  Arms: Group A
Biological: Normal saline injection — All subjects of this group will receive 2 sessions of normal saline penile injection with 30 +/- 3 day treatment interval for all subjects, 10 ml of normal saline will be injected at each session.
  Arms: Group B

SUMMARY:
The primary objective of the present study is to investigate and compare the treatment efficacy of PRP injection vs placebo treatment in men with mild-moderate vasculogenic ED, as measured by IIEF.The secondary objective of the present clinical trial is to study the adverse events and safety of the PRP injection treatment in vasculogenic ED patients

ELIGIBILITY:
Inclusion Criteria:

1. Consent to participate.
2. Age 40-70 years.
3. Sexually active in a stable, heterosexual relationship of more than three months duration.
4. Presence of Erectile Dysfunction for at least 6 months.
5. IIEF-ED: 11-25 at visit 1
6. PDE5i users and report some/good response to PDE5i at the last month before screening.
7. Agree to suspend all ED therapy for the duration of the study.
8. Agree to attempt sexual intercourse at least 4 times every 4 weeks, for the duration of the study without being under the influence of alcohol or recreational drugs. Agree to document the outcome using the Sexual Encounter Profile (SEP) diary, as needed.

Exclusion Criteria:

1. Previous major pelvic surgery or pelvic trauma that could impact erectile function, such as radical prostatectomy, radical cystectomy, rectal surgery. Patients with previous TURP surgery without sequelae of iatrogenic ED, may be included.
2. Previous penile surgery of any kind except circumcision and condyloma removal, such as penile lengthening, penile cancer surgery, penile plication, grafting.
3. Previous history of priapism or penile fracture
4. Previous radiation therapy to pelvis.
5. Abnormal morning serum testosterone level defined as a value lower than 300 ng/dL +/- 5 %(indicative of untreated hypogonadism), or greater than 1197 ng/dL +/- 5%.
6. Current or previous hormone usage, other than prescribed testosterone, clomiphene or thyroid medication. Subjects with prior or current use of hormonal treatment for prostate cancer are also excluded.
7. Psychogenic ED.
8. Peyronie's Disease or penile curvature that negatively influences sexual activity.
9. Anatomical or neurological abnormalities in the treatment area.
10. Any untreated medical condition (medical history)
11. Patients with generalized polyneuropathy, or neurological conditions irrespective of cause, such as severe diabetes, multiple sclerosis or Parkinson's Disease.
12. Refusal to suspend ED therapy for duration of study. Subjects who are using Tadalafil as a treatment for BPH (Benign Prostatic Hyperplasia) will also be excluded.
13. Men deemed not healthy enough to participate in sexual activity.
14. Any condition or behavior that indicates to the Principal Investigator that the subject is unlikely to be compliant with study procedures and visits.
15. Any health history or laboratory result that indicates to the Principal Investigator that the subject has a significant medical condition and should not participate in the study.
16. History of consistent treatment failure with PDE5 inhibitors for therapy of ED.
17. Any history of significant psychiatric disease, such as bipolar disorder or psychosis, greater than one lifetime episode of major depression, current depression of moderate or greater severity. Patients who are currently using SSRI or psychotropic medications.
18. Partners who are < 18 years of age, who are nursing, who are known to be pregnant at screening, who wish to become pregnant during the study period, who have any gynecologic problems, sexual dysfunction, or major medical conditions that would limit participation in sexual intercourse.
19. Patients with any hematological disorder.

Ages: 40 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 60 (Actual)
Dates: Start 2019-09-02 (Actual); Primary Completion 2020-03-26 (Actual); Study Completion 2020-09-24 (Actual)

PRIMARY OUTCOMES:
The % of patients in each group who attain Minimal Clinically Important Difference (MCID) in International Index of Erectile Function -Erectile Function (IIEF-EF) domain from baseline to 24 weeks after final treatment. | at 24 weeks follow up visit
  MCID is defined according to baseline ED severity as:Improvement by 5 or more in the EF domain score of the IIEF for patients with moderate ED at baseline and by 2 or more in the EF domain score of the IIEF for patients with moderate ED at baseline

SECONDARY OUTCOMES:
The % of patients in each group who attain MCID in IIEF-EF domain from baseline to 12 weeks after final treatment. | at 12 weeks follow up visit
  MCID is defined according to baseline ED severity as:Improvement by 5 or more in the EF domain score of the IIEF for patients with moderate ED at baseline and by 2 or more in the EF domain score of the IIEF for patients with moderate ED at baseline
The % of patients in each group who attain MCID in IIEF-EF domain from baseline to 4 weeks after final treatment. | at 4 weeks follow up visit
  MCID is defined according to baseline ED severity as:Improvement by 5 or more in the EF domain score of the IIEF for patients with moderate ED at baseline and by 2 or more in the EF domain score of the IIEF for patients with moderate ED at baseline
The difference between the PRP group (2 sessions of PRP) and the placebo group in the change of the IIEF-ED score from baseline to 4 weeks after final treatment. | baseline and 4 weeks follow up visit
  EF domain of the IIEF questionnaire will be completed. IIEF-EF consists of items 1,2,3,4,5,15 of the IIEF questionnaire.According to the score of the iIEF-EF there are five categories of erectile function: 1-10 (Severe Erectile Dysfunction), 11-16(Moderate dysfunction), 17-21(Mild to moderate dysfunction), 22-25(Mild dysfunction), 26-30 (No dysfunction).
The difference between the PRP group (2 sessions of PRP) and the placebo group in the change of the IIEF-ED score from baseline to 12 weeks after final treatment. | baseline and 12 weeks follow up visit
  EF domain of the IIEF questionnaire will be completed.IIEF-EF consists of items 1,2,3,4,5,15 of the IIEF questionnaire.According to the score of the iIEF-EF there are five categories of erectile function: 1-10 (Severe Erectile Dysfunction), 11-16(Moderate dysfunction), 17-21(Mild to moderate dysfunction), 22-25(Mild dysfunction), 26-30 (No dysfunction)
The difference between the PRP group (2 sessions of PRP) and the placebo group in the change of the IIEF-ED score from baseline to 24 weeks after final treatment. | baseline and 24 weeks follow up visit
  EF domain of the IIEF questionnaire will be completed.IIEF-EF consists of items 1,2,3,4,5,15 of the IIEF questionnaire.According to the score of the iIEF-EF there are five categories of erectile function: 1-10 (Severe Erectile Dysfunction), 11-16(Moderate dysfunction), 17-21(Mild to moderate dysfunction), 22-25(Mild dysfunction), 26-30 (No dysfunction)
The difference between the PRP group (2 sessions of PRP) and the placebo group in the change in Sexual Encounter Profile Question 3 (SEP3) score from baseline to 4 weeks after final treatment. | baseline and 4 weeks follow up visit
  The percent of subjects who answer ''YES'' in question 3 of SEP questionnaire will be reported
The difference between the PRP group (2 sessions of PRP) and the placebo group in the change in Sexual Encounter Profile Question 3 (SEP3) score from baseline to 12 weeks after final treatment. | baseline and 12 weeks follow up visit
  The percent of subjects who answer ''YES'' in question 3 of SEP questionnaire will be reported
The difference between the PRP group (2 sessions of PRP) and the placebo group in the change in Sexual Encounter Profile Question 3 (SEP3) score from baseline to 24 weeks after final treatment. | baseline and 24 weeks follow up visit
  The percent of subjects who answer ''YES'' in question 3 of SEP questionnaire will be reported
The difference between the PRP group (2 sessions of PRP) and the placebo group in Erectile Dysfunction Inventory of Treatment Satisfaction (EDITS) questionnaire score | 4,12, 24 weeks follow up visit
  EDITS is an 11-item validated questionnaire assessing treatment satisfaction. The 11 items in the EDITS questionnaire are combined into an index score by computing the mean of the 11 item scores and multiplying this value by 25. This results in an EDITS index score with a range of 0 (extremely low treatment satisfaction) to 100 (extremely high treatment satisfaction) for an individual patient.
The difference between the PRP group (2 sessions of PRP) and the placebo group in the the Pain Visual Analogue Scale (VAS) after each injection treatment session | at week 0 and 4
  It will be assessed by the pain VAS, right after each LIST session. Pain VAS is a unidimensional measure of pain intensity . It is a continuous scale comprised of a horizontal (HVAS) or vertical (VVAS) line, usually 10 centimeters (100 mm) in length, anchored by 2 verbal descriptors, one for each symptom extreme. For pain intensity, the scale is most commonly anchored by "no pain" (score of 0) and "pain as bad as it could be" or "worst imaginable pain" (score of 100 [100-mm scale]. To avoid clustering of scores around a preferred numeric value, numbers or verbal descriptors at intermediate points are not recommended. The following cut points on the pain VAS have been recommended: no pain (0-4 mm), mild pain (5-44 mm), moderate pain (45-74 mm), and severe pain (75- 100 mm
Number of patients with treatment related adverse events | 28 weeks
  Potential treatment related adverse events after the first PRP injection session and during the 3 month follow up period will be reported

CONTACTS AND LOCATIONS:
Overall Officials: Dimitrios Hatzichristou, Prof., Principal Investigator — G.Gennimatas General Hospital, Thessaloniki,Greece
Locations (1):
- G.Gennimatas Hospital, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Epifanova MV, Gvasalia BR, Durashov MA, Artemenko SA. Platelet-Rich Plasma Therapy for Male Sexual Dysfunction: Myth or Reality? Sex Med Rev. 2020 Jan;8(1):106-113. doi: 10.1016/j.sxmr.2019.02.002. Epub 2019 Mar 19. PMID 30898594
- [Background] Scott S, Roberts M, Chung E. Platelet-Rich Plasma and Treatment of Erectile Dysfunction: Critical Review of Literature and Global Trends in Platelet-Rich Plasma Clinics. Sex Med Rev. 2019 Apr;7(2):306-312. doi: 10.1016/j.sxmr.2018.12.006. Epub 2019 Mar 2. PMID 30833169
- [Background] Wu YN, Wu CC, Sheu MT, Chen KC, Ho HO, Chiang HS. Optimization of platelet-rich plasma and its effects on the recovery of erectile function after bilateral cavernous nerve injury in a rat model. J Tissue Eng Regen Med. 2016 Oct;10(10):E294-E304. doi: 10.1002/term.1806. Epub 2013 Aug 16. PMID 23950105